CLINICAL TRIAL: NCT05046119
Title: Factors Associated With Migraine Refractoriness to Preventive Treatments: Psychological Aspects and Relationship With Components of the Endocannabinoid System
Brief Title: Psychological and Biological Markers of Refractory Migraine
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ReMi2021
Record Dates: First submitted 2021-09-02; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Migraine
Keywords: Migraine; Refractoriness; Monoclonal antibodies directed against CGRP; Psychological disturbances; Endocannabinoid system
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A sample of peripheral blood (30ml) for the evaluation of gene expression of enzymes involved in the synthesis (arachidonoylphospatidylethanolamine phospholipase D (NAPE-PLD) and diacylglycerol lipase α (DAGL-α)) and degradation (Fatty acid amide hydrolase (FAAH) or monoacylglycerol lipase (MAGL)) of endocannabinoids and their receptors (CB1 and CB2) in peripheral mononuclear cells (PBMC), through rtPCR method. In addition, in the same subjects we will evaluate plasma levels of AEA and its congener Palmitoylethanolamide, known to be altered in chronic migraine. The outcomes at 3 and 6 months will be analyzed cross-sectionally.
Oversight: Data Monitoring Committee: No

SUMMARY:
The term "refractory" migraine describes a particularly aggressive form of the disease in which the patient does not benefit from any of the preventive therapies with the various classes of drugs available, including treatment with monoclonal antibodies directed against Calcitonin Gene Related Peptide (CGRP).

Anxiety, depressive symptoms, somatization, and pain hypersensitivity are significantly more prevalent in refractory migraineurs than in non-refractory subjects who benefit from preventive therapies, suggesting that these symptoms may contribute to treatment refractoriness. Recently, in a preliminary study on the efficacy of a CGRP-targeting monoclonal antibody in Chronic Migraine (CM) patients with at least 3 failures to previous preventive treatments, the investigators showed a higher prevalence of psychological disturbances in those who did respond to the monoclonal antibody compared with the responders. These data, although preliminary, point to a more psychologically complicated picture in non-responder patients compared with responders. To date, however, no neurobiological evaluations are available to explain how psychological comorbidities may contribute to treatment refractoriness. Isolated clinical evidence and growing pre-clinical evidence suggests a role for the endocannabinoid system in migraine. Hence, the present study aims to identify psychological and biological factors associated with refractory migraine. The investigators' hypothesis is that patients presenting with psychological disorders may bear an associated dysfunction of the endocannabinoid system, which makes them more resistant to migraine preventive therapies, including monoclonal antibodies directed against CGRP.

DETAILED DESCRIPTION:
Migraine is a common and highly disabling condition, representing the second-leading cause of disability in the global ranking of most disabling diseases . In the majority of individuals, the disease manifests as episodic (EM), with attacks recurring weekly or monthly. In a smaller (2-3% of the general population), but still significant portion of patients, migraine becomes chronic, i.e., occurring on at least 15 days per month (CM).

Previous studies have shown that CM patients are characterized by the presence of multiple psychiatric comorbidities compared with subjects with episodic migraine and healthy controls. In recent years, it has also been shown that among the neurobiological systems involved in the genesis and development of mental disorders, the endocannabinoid system (ES) appears to play an active role. In particular, patients with these disorders are characterized, at the level of peripheral cells, by a gene alteration of cannabinoid receptors.

Several studies reported the involvement of SE in immune responses, psychological processes, transduction of neurobiological signals and pain, including migraine pain. Recently it has been shown that the peripheral gene expression of enzymes involved in the metabolism of anandamide (AEA) and 2-aciglycerol (2-AG), the two best known endocannabinoids, is altered in migraine patients, but more markedly in the chronic subtype, suggesting a role for these lipid molecules not only in the pathophysiology of the disease, but also in its exacerbation. The role of CGRP in the pathophysiology of migraine has now been demonstrated, although the mechanism of action at both peripheral and central levels and its possible interactions with other pathways are not completely known.

The term "refractory" migraine describes a particularly aggressive form of the disease in which the patient does not benefit from any of the preventive therapies with the various classes of drugs available, including treatment with monoclonal antibodies directed against CGRP (Consensus document of the European Headache Federation).

Anxiety, depressive symptoms, somatization, and pain hypersensitivity are significantly more prevalent in refractory migraineurs than in non-refractory subjects who benefit from preventive therapies, suggesting that these symptoms may contribute to treatment refractoriness. Recently, in a preliminary study regarding the efficacy of monoclonal antibody targeting CGRP in CM patients refractory to at least three preventive therapies,the investigators showed a higher prevalence of personality disorders (77% vs 37%) in those who were not responding to treatment at 1 year (non-responders: reduction in migraine days <50%), compared with those who were responding (responders: reduction in migraine days ≥50%). Non-responders were also characterized by a higher prevalence of anxiety spectrum disorders and more stressful events than responders. These data, although preliminary, point to a more psychologically complicated picture in non-responder patients compared with responders. To date, however, no neurobiological data are available to explain how psychological comorbidities may contribute to treatment refractoriness.

In this frame, the present study aims to identify psychological and potential biochemical/molecular factors associated with refractory migraine. The investigators' hypothesis is that patients presenting with psychological disorders may bear an associated dysfunction of the endocannabinoid system, which makes them more resistant to migraine preventive therapies, including monoclonal antibodies directed against CGRP.

There will be a screening phase of one month in which patients will complete a daily headache diary in which they will note the occurrence, intensity and duration of attacks, as well as the use of symptomatic drugs. At baseline patients will undergo the psychological and biochemical/molecular evaluation. Subjects will then be treated with one of the three commercially available monoclonal antibodies targeting CGRP and will continue to record the characteristics of attacks and the use of symptomatic drugs in their headache diary. Follow-up visits are foreseen after 3 and 6 months of treatment. At 6 months, patients will be divided into 2 groups (responder or not responder to the treatment) depending on the reduction of monthly migraine days in the previous 3 months (>50% and <50%, respectively).

The patients who failed to respond to the treatment will be considered refractory.

Psychological evaluation: All patients will be evaluated by psychological interview and by adopting the DSM-V criteria for personality disturbances, anxiety and mood disorders. All patients will also be administered the Hospital Anxiety and Depression Scale (HADS) the Toronto Alexithymia Scale 20 (TAS-20), severity of dependence questionnaires (Severity Dependence Scale - SDS - and Leeds Dependence Questionnaire - LDQ), questionnaires related to Childhood trauma and Stressful life events.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical characteristics that meet the criteria of the current International Headache Classification for Migraine or Chronic Migraine.
2. Age >18, <65 years of both sexes
3. At least 8 days of migraine/month and Migraine Disability Assessment Questionnaire (MIDAS) score greater than 11 at baseline*.
4. Lack of benefit or intolerance or contraindication to at least three classes of drugs for the preventive therapy of migraine*.

   * Drug Italian Agency (AIFA) criteria for the prescription of monoclonal antibodies directed against CGRP.

Exclusion Criteria:

1. dementia, psychosis, mental retardation
2. women of childbearing age without contraceptive protection, pregnant and lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eighty participants with EM and CM will be recruited at the Headache Science and Neurorehabilitation Centre of the IRCCS Mondino Foundation. The diagnosis of EM and CM is formulated according to the guidelines of the ICHD-III version (EM or CM with previous failure to at least 3 of the following classes of antimigraine preventive drugs :beta-blockers, antidepressants, calcium antagonists and, for CM, onabotulinumtoxinA).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-09-15 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Personality disorders | Change from baseline to 3-month to 6-month
  To evaluate the association of refractory migraine with personality disorders (according to Diagnostic and Statistical Manual of mental disorders - DSM V criteria) in subjects with resistant migraine undergoing therapy with monoclonal antibodies directed against CGRP.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Baseline, pre-receiving the treatment
  The HADS is a fourteen item scale that generates: seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3. Higher scores are worst outcomes
Toronto Alexitimia Scale 20 (TAS-20) | Baseline, pre-receiving the treatment
  The TAS is a 20-item instrument that is one of the most commonly used measures of alexithymia. The TAS-20 uses cutoff scoring: equal to or less than 51 = non-alexithymia, equal to or greater than 61 = alexithymia. Scores of 52 to 60 = possible alexithymia.
Childhood traumas questionnaire | Baseline, pre-receiving the treatment
  The Childhood Trauma Questionnaire (CTQ) is a retrospective, self-report measure that was developed to provide a brief, reliable, and valid assessment of a broad range of traumatic experiences in childhood. It contains 70 items arranged according to four factors: physical and emotional abuse, emotional neglect, sexual abuse, and physical neglect. Responses are quantified on a 5-point Likert-type scale according to the frequency with which experiences occurred, with 1 = "never true" and 5 = "very often true.
Stressful life events questionnaire (SLESQ) | Baseline, pre-receiving the treatment
  SLESQ is a 13-item self-report measure for non-treatment seeking samples that assesses lifetime exposure to traumatic events. Eleven specific and two general categories of events, such as a life-threatening accident, physical and sexual abuse, witness to another person being killed or assaulted, are examined. For each event, respondents are asked to indicate whether the event occurred ("yes" or "no"), their age at time of the event, as well as other specific items related to the event, such as the frequency, duration, whether anyone died, or was hospitalization, etc.
The Leeds Dependence Questionnaire (LDQ) | Baseline, pre-receiving the treatment
  The LDQ has been developed as part of a treatment evaluation package. The LDQ is a 10-item, self completion questionnaire designed to measure dependence upon a variety of substances. All items are scored 0-1-2-3.
Severity of Dependence Scale (SDS) | Baseline, pre-receiving the treatment
  The Severity of Dependence Scale (SDS) is a 5-item self-administered questionnaire that provides a score indicating the severity of dependence on drugs. Higher scores are worst outcomes
Endocannabinoid System (ES) | Baseline, pre-receiving the treatment
  Main components of the ES at the peripheral level

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Tassorelli, Prof, Principal Investigator — Headache Science Center
Locations (1):
- Headache Science Center, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ashton CH, Moore PB. Endocannabinoid system dysfunction in mood and related disorders. Acta Psychiatr Scand. 2011 Oct;124(4):250-61. doi: 10.1111/j.1600-0447.2011.01687.x. Epub 2011 Mar 9. PMID 21916860
- [Background] Bottiroli S, Galli F, Viana M, De Icco R, Bitetto V, Allena M, Pazzi S, Sances G, Tassorelli C. Negative Short-Term Outcome of Detoxification Therapy in Chronic Migraine With Medication Overuse Headache: Role for Early Life Traumatic Experiences and Recent Stressful Events. Front Neurol. 2019 Mar 7;10:173. doi: 10.3389/fneur.2019.00173. eCollection 2019. PMID 30899242
- [Background] Bottiroli S, Galli F, Viana M, Sances G, Tassorelli C. Traumatic Experiences, Stressful Events, and Alexithymia in Chronic Migraine With Medication Overuse. Front Psychol. 2018 May 14;9:704. doi: 10.3389/fpsyg.2018.00704. eCollection 2018. PMID 29867669
- [Background] Bottiroli S, Viana M, Sances G, Ghiotto N, Guaschino E, Galli F, Vegni E, Pazzi S, Nappi G, Tassorelli C. Psychological factors associated with failure of detoxification treatment in chronic headache associated with medication overuse. Cephalalgia. 2016 Dec;36(14):1356-1365. doi: 10.1177/0333102416631960. Epub 2016 Feb 15. PMID 26879321
- [Background] Cupini LM, Bari M, Battista N, Argiro G, Finazzi-Agro A, Calabresi P, Maccarrone M. Biochemical changes in endocannabinoid system are expressed in platelets of female but not male migraineurs. Cephalalgia. 2006 Mar;26(3):277-81. doi: 10.1111/j.1468-2982.2005.01031.x. PMID 16472333
- [Background] Cupini LM, Costa C, Sarchielli P, Bari M, Battista N, Eusebi P, Calabresi P, Maccarrone M. Degradation of endocannabinoids in chronic migraine and medication overuse headache. Neurobiol Dis. 2008 May;30(2):186-9. doi: 10.1016/j.nbd.2008.01.003. Epub 2008 Feb 1. PMID 18358734
- [Background] De Icco R, Greco R, Demartini C, Vergobbi P, Zanaboni A, Tumelero E, Reggiani A, Realini N, Sances G, Grillo V, Allena M, Tassorelli C. Spinal nociceptive sensitization and plasma palmitoylethanolamide levels during experimentally induced migraine attacks. Pain. 2021 Sep 1;162(9):2376-2385. doi: 10.1097/j.pain.0000000000002223. PMID 33587406
- [Background] Iani L, Lauriola M, Costantini M. A confirmatory bifactor analysis of the Hospital Anxiety and Depression Scale in an Italian community sample. Health Qual Life Outcomes. 2014 Jun 5;12:84. doi: 10.1186/1477-7525-12-84. PMID 24902622
- [Background] Ibarra-Lecue I, Pilar-Cuellar F, Muguruza C, Florensa-Zanuy E, Diaz A, Uriguen L, Castro E, Pazos A, Callado LF. The endocannabinoid system in mental disorders: Evidence from human brain studies. Biochem Pharmacol. 2018 Nov;157:97-107. doi: 10.1016/j.bcp.2018.07.009. Epub 2018 Jul 17. PMID 30026022
- [Background] Sacco S, Braschinsky M, Ducros A, Lampl C, Little P, van den Brink AM, Pozo-Rosich P, Reuter U, de la Torre ER, Sanchez Del Rio M, Sinclair AJ, Katsarava Z, Martelletti P. European headache federation consensus on the definition of resistant and refractory migraine : Developed with the endorsement of the European Migraine & Headache Alliance (EMHA). J Headache Pain. 2020 Jun 16;21(1):76. doi: 10.1186/s10194-020-01130-5. PMID 32546227
- [Background] Sarchielli P, Pini LA, Coppola F, Rossi C, Baldi A, Mancini ML, Calabresi P. Endocannabinoids in chronic migraine: CSF findings suggest a system failure. Neuropsychopharmacology. 2007 Jun;32(6):1384-90. doi: 10.1038/sj.npp.1301246. Epub 2006 Nov 22. PMID 17119542
- [Background] Tassorelli C, Greco R, Silberstein SD. The endocannabinoid system in migraine: from bench to pharmacy and back. Curr Opin Neurol. 2019 Jun;32(3):405-412. doi: 10.1097/WCO.0000000000000688. PMID 30883435
- [Background] Viana M, Bottiroli S, Sances G, Ghiotto N, Allena M, Guaschino E, Nappi G, Tassorelli C. Factors associated to chronic migraine with medication overuse: A cross-sectional study. Cephalalgia. 2018 Dec;38(14):2045-2057. doi: 10.1177/0333102418761047. Epub 2018 Apr 10. PMID 29635935